CLINICAL TRIAL: NCT05378789
Title: Appropriation and Impact of the Introduction of Naps During Night Work by Intensive Care Caregiver - One Year Review
Acronym: MARIENAIE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Departemental Vendee (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CHD21_0119
Record Dates: First submitted 2022-05-13; First posted 2022-05-18 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Nap
Keywords: nap; ICU; nurse; Shift work

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 20-min nap (Experimental): ICU nurses can take a 20-minute nap between 2 and 5 am according to a rotation of personal.
  Naps will be carried out with the help of a Nap and Up ® cocoon deckchair.
  Interventions: Procedure: Nap

INTERVENTIONS:
Procedure: Nap — ICU nurses can take a 20-mn nap between 2 and 5 am according to a rotation of personal.
  Naps will be carried out with the help of a Nap and Up ® cocoon deckchair.

SUMMARY:
MARIENAIE study is a pilot study on the feasibility and appropriation of nocturnal naps by a team of paramedical caregivers alternating a 12-hour day/night work rhythm for a period of 1 year. To date no study on the impact of nap in ICU on a long period was published.

This study will also explore : the factors favouring or hindering the implementation of this strategy and its maintenance over time through a concomitant sociological qualitative study, the evolution over time of the parameters of perceived nocturnal sleepiness and the immediate impact of the realization of naps on this sleepiness and the evolution over time of the medium-term impact with the help of questionnaires exploring various dimensions concerning the working conditions and health (somatic health, stress, psychosocial risks, evaluation of the working environment).

ELIGIBILITY:
Inclusion Criteria:

* Paramedic working 12 hours alternating day and night in the ICU department of the Vendee departmental hospital center.

Exclusion Criteria:

* Pregnant woman.
* Caregiver with knowledge of a scheduled departure from the ICU within 2 months after the start of the project.
* Caregiver refusing to participate in the project.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2022-05-30 (Actual); Primary Completion 2023-07-15 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Nap appropriation | 12 months after baseline
  Proportion of the number of nights worked with micro-naps to the number of nights worked by a caregiver over a year.

CONTACTS AND LOCATIONS:
Overall Officials: Mélanie ROUGIER, Principal Investigator — Centre hospitalier departemental Vendée
Locations (1):
- Centre hospitalier départemental Vendee, La Roche-sur-Yon, France

IPD SHARING:
Plan to Share IPD: No